CLINICAL TRIAL: NCT03470168
Title: Hyperbaric Oxygenation in Treatment of Alcohol Dependence Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Collaborators: INCRE fellowship from DBT, govt of India (Unknown)
Responsible Party: Principal Investigator, Dr Geomy George Chakkalakkudy, Assistant Professor, Department of Psychiatry, Jubilee Mission Medical College and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 25/16/IEC/JMMC&RI
Record Dates: First submitted 2017-03-02; First posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Alcohol Withdrawal Symptoms; Delirium Tremens (DTs)
MeSH Terms: conditions — Alcohol Withdrawal Delirium | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: 30 alcohol dependent patients were divided into A: Treatment group and B: Placebo group using simple randomization technique.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperbaric Oxygen Therapy (Experimental): Received the Hyperbaric Oxygen therapy treatment at 2.4 ATA for 90 minutes each day.
  Interventions: Device: Hyperbaric Oxygenation Therapy
- Placebo group (Placebo Comparator): were also taken inside the Hyperbaric Chamber, but received only normobaric oxygen therapy for the same period of time at 1 ATA
  Interventions: Device: Normobaric Oxygenation therapy

INTERVENTIONS:
Device: Hyperbaric Oxygenation Therapy — Received the Hyperbaric Oxygen therapy treatment at 2.4 ATA for 90 minutes each day.
  Other Names: Treatment group
  Arms: Hyperbaric Oxygen Therapy
Device: Normobaric Oxygenation therapy — Received the Normobaric Oxygen therapy treatment at 1 ATA for 90 minutes each day.
  Other Names: Placebo group
  Arms: Placebo group

SUMMARY:
A 30 alcohol dependent patients were divided into A: Treatment group and B: Placebo group using simple randomization technique. (Liver function tests) GGT, ALT and AST levels and MCV (Mean corpuscular volume) at admission and 2 weeks later were estimated. Daily withdrawal symptoms were assessed using the Clinical Institute Withdrawal Assessment scale (CIWA-Ar) and DTs by Delirium Observation Screening (DOS) Scale (version 0 - 1). The data collected from the two groups were compared.

DETAILED DESCRIPTION:
This is a prospective randomized study conducted in the de-addiction ward of department of Psychiatry, Jubilee Mission Medical College, Thrissur, Kerala. The study period was from 16/11/2014 to 30/04/2016 (17 months and 14 days). This study was approved by the Institutional Review Board. Male patients aged between 20-60 years with alcohol dependence as per ICD-10 criteria, who presented with AWS and DTs on admission or during the course in our ward were recruited to the study. Those patients suffering from severe physical illness incapacitating for psychiatric evaluation, who are mentally retarded, who have primary psychiatric disorders like psychosis, mood disorder and those with neurodegenerative disorders like Dementia, Cerebrovascular accidents were excluded. In each case the patient and relatives were explained about the purpose of the study, its nature and the possible advantages and disadvantages of taking part in the study. An informed consent for the study was obtained from the patient as well as the relatives. Each subject was evaluated by a proper history, general examination, systemic examination, detailed mental status examination, laboratory investigations and psychometric evaluation (if needed) at the time of admission. The intended laboratory investigations were γ-glutamyl transferase (GGT), Alanine aminotranferease (ALT), aspartate aminotransferase (AST) and MCV (mean corpuscular volume of RBCs). These were done at time of recruitment. The severity of withdrawal symptoms was assessed using the Clinical Institute Withdrawal Assessment scale (CIWA-Ar) and that for delirium was rated using the Delirium Observation Screening (DOS) Scale (version 0 - 1). All patients had an ECG and a baseline echocardiography to assess their cardiac status. The echocardiography was repeated at the end of 2 weeks. Parameters to be studied included ejection fraction, and end systolic residual volume. All the patients had an ENT consultation to rule out any tympanic membrane pathologies.

The total of 30 patients divided to A: Treatment group and B: Control using Simple randomization technique using random number generating software (ver. 1). A, received the Hyperbaric Oxygen therapy treatment at 2.4 ATA for 90 minutes each day. B were also taken inside the Hyperbaric Chamber, but received only normobaric oxygen therapy for the same period of time at 1 ATA. All of the cases received all standard medications. Hyperbaric oxygenation was done at our hospital in a monoplace chamber (Oxicab,HyperbaricSAC, Peru). The entire session was carried out in presence of the Hyperbaric Physician and technician. Prior to this therapy the documentation of pulse rate, Blood Pressure and Blood sugar were done as standard procedure. The Hyperbaric sessions were done for 10 days in a row one time daily. Daily general examination, systemic examination, detailed mental status examination and administration of CIWA scale and DOS scale were carried out till the day of discharge.

Laboratory investigations were repeated after two weeks. The patients were discharged when the biological functions were adequate, physical and mental conditions were stable and when they were motivated to remain abstinent from alcohol. Parameters assessed in two groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged between 20-60 years with alcohol dependence as per ICD-10 criteria, who presented with AWS and DTs on admission or during the course in our ward were recruited to the study.

Exclusion Criteria:

* Those patients suffering from severe physical illness incapacitating for psychiatric evaluation, who are mentally retarded, who have primary psychiatric disorders like psychosis, mood disorder and those with neurodegenerative disorders like Dementia, Cerebrovascular accidents were excluded.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Rate of improvement | 1 year
  faster recovery from DTs and withdrawal symptoms.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sassi,F.(ed.), Tackling Harmful Alcohol Use: Economics and Public Health Policy, OECD Publishing, Paris 2015.
- [Background] World Health Organization (WHO) -Global Status report on Alcohol and Health -2014
- [Background] American psychiatric association; Diagnostic and statistical manual of mental disorders; 4th edition; Text Revision (DSM IV TR)
- [Background] Caetano R, Clark CL, Greenfield TK. Prevalence, trends, and incidence of alcohol withdrawal symptoms: analysis of general population and clinical samples. Alcohol Health Res World. 1998;22(1):73-9. PMID 15706737